CLINICAL TRIAL: NCT04835181
Title: Electroacupuncture Combined With Umbilical Moxibustion on Abdominal Obesity of Yang Deficiency: A Study Protocol for a Randomized Controlled Trial
Brief Title: Electroacupuncture Combined With Umbilical Moxibustion on Abdominal Obesity of Yang Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBPCIC-2020-05
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture combined with umbilical moxibustion (Experimental)
  Interventions: Behavioral: Electroacupuncture combined with umbilical moxibustion
- Electroacupuncture (Active Comparator)
  Interventions: Behavioral: Electroacupuncture

INTERVENTIONS:
Behavioral: Electroacupuncture combined with umbilical moxibustion — ①Umbilical moxibustion intervention: point selection: Shenque point Operation: Place the aconite cake on the Shenque point, place the Aizhu in the middle of the aconite cake, ignite the Aizhu and apply moxibustion to make the local warm sensation without burning pain, until the skin is flushed.
  ②Electro-acupuncture intervention: Acupoint selection: Tianshu, Zusanli, Zhongwan, Moisture, Daheng, Vein, Waterway, Huaroumen, Abdominal Knot.
  Operation: supine position, routine skin disinfection. After routine acupuncture at the acupoints, apply the technique of flattening, replenishing, relieving, and relieving qi. Tianshu and Daheng points, respectively, were horizontally connected to the electrodes of the electroacupuncture instrument on the needle handles of the bilateral Tianshu and Daheng points.
  Electroacupuncture parameters: density wave, current intensity 1-5mA, electroacupuncture intensity is subject to patient tolerance.
  Arms: Electroacupuncture combined with umbilical moxibustion
Behavioral: Electroacupuncture — ②Electro-acupuncture intervention: Acupoint selection: Tianshu, Zusanli, Zhongwan, Moisture, Daheng, Vein, Waterway, Huaroumen, Abdominal Knot.
  Operation: supine position, routine skin disinfection. After routine acupuncture at the acupoints, apply the technique of flattening, replenishing, relieving, and relieving qi. Tianshu and Daheng points, respectively, were horizontally connected to the electrodes of the electroacupuncture instrument on the needle handles of the bilateral Tianshu and Daheng points.
  Electroacupuncture parameters: density wave, current intensity 1-5mA, electroacupuncture intensity is subject to patient tolerance.
  Arms: Electroacupuncture

SUMMARY:
Obesity is a chronic metabolic disease that seriously harms human health, while abdominal obesity is more closely related to diseases such as type 2 diabetes, cardiovascular disease, and tumors, and has a higher risk. In recent years, traditional Chinese medicine therapy has become the choice of more and more obese patients, and acupuncture therapy is also known as a green therapy for weight loss due to its safety and no side effects. Through the analysis of the TCM physique types of obese people, it is found that Yang-deficiency constitution is one of the TCM constitution types closely related to simple obesity. This topic is based on the constitution theory of traditional Chinese medicine, and on the basis of the earlier research that has clarified the weight loss and lipid-lowering effects of electroacupuncture, it further aims at the type of yang deficiency in obese people, and clarifies the regulation and improvement of umbilical moxibustion on the constitution of obese patients with yang deficiency. In this project, patients with abdominal obesity with yang-deficiency constitution were divided into electro-acupuncture + umbilical moxibustion group and electro-acupuncture group to observe and analyze the advantages and effects of electro-acupuncture combined with umbilical moxibustion on the improvement of obesity symptoms and physical fitness of patients. The ELISA method was used to determine the metabolic indexes related to yang-deficiency constitution, to further clarify the material basis of electroacupuncture combined with umbilical moxibustion to improve the yang-deficiency constitution of patients with abdominal obesity, and to provide scientific and reasonable theoretical guidance for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. People who meet the following diagnostic criteria and are diagnosed with abdominal obesity due to yang deficiency:

1. Diagnostic criteria for abdominal obesity: Refer to the criteria in the "Guidelines for the Comprehensive Medical Management of Obese People" jointly issued by the American Academy of Clinical Endocrinologists (AACE) and the American College of Endocrinology (ACE) in May 2016: male waist circumference ≥85cm, female Waist circumference ≥80cm can be diagnosed as abdominal obesity.
2. Yang Deficiency Quality Criteria: Meet the diagnostic criteria of Yang Deficiency in the "Classification and Judgment Table of Traditional Chinese Medicine Constitution". Common manifestations are chills, cold limbs, swollen face, pale complexion, pale tongue, white slippery fur, and weak pulse.

2. Age: 18 to 55 years old; 3. Sign the informed consent and voluntarily accept the intervention method of this project.

Exclusion Criteria:

1. Severe lung, heart, liver, kidney and other diseases;
2. Combined endocrine diseases (polycystic ovary syndrome, hypothyroidism, Cushing syndrome, etc.);
3. Have a history of surgery to lose weight; have a history of adhesions after previous surgery;
4. Have taken drugs that are known to affect weight or appetite in the past 3 months, such as weight loss drugs, corticosteroids, etc.; have used hormone drugs, lipid-lowering drugs, and hypoglycemic drugs in the past 3 months;
5. Women during pregnancy, lactation and menopause;
6. Participated in clinical research on weight loss in the past 3 months; Those who meet any of the above will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Waist circumference(WC) at week 12 | Baseline and Week 12
  The horizontal girth through the center of the umbilicus

SECONDARY OUTCOMES:
Weight(WG) | Week 0, Week 4, Week 8, Week 12
  Weight(WG) will be measured.
BMI(weight/(height) | Week 0, Week 4, Week 8, Week 12
  BMI (weight/(height) will be measured.
hip circumference(HC) | Week 0, Week 4, Week 8, Week 12
  hip circumference(HC) will be measured.
Waist-to-hip ratio(waist circumference/hip circumference) | Week 0, Week 4, Week 8, Week 12
  waist-to-hip ratio(waist circumference/hip circumference) will be measured.
The impact of weight on quality of life (IWQOL)-Lite scale | Week 0, Week 4, Week 8, Week 12
  The impact of weight on quality of life (IWQOL)- Lite scale will be measured to assess the improvement in the quality of life of participants. The minimum value is 31，the maximum value is 155. The lower the total score, the lighter the clinical symptoms of the patient.
The 10-item Kessler Psychological Distress (K10) Scale | Week 0, Week 4, Week 8, Week 12
  The 10-item Kessler Psychological Distress (K10) Scale will be measured to assess participant's mental state. The minimum value is 10，the maximum value is 50. The lower the total score, the lighter the clinical symptoms of the patient.
TCM Physique Classification and Judgment Table | Week 0, Week 4, Week 8, Week 12
  Refer to the physical characteristics in the "Traditional Chinese Medicine Physique Classification and Judgment Table" to determine the changes in the yang deficiency constitution of the participants. The symptom score is quantified in 5 levels: always, 5 points; often, 4 points; sometimes, 3 points; very Less, 2 points, no, 1 point. Then calculate the constitutional symptom conversion score, and the change value of the constitutional symptom conversion score compared with the baseline.The minimum value is 0，the maximum value is 100. The lower the total score, the lighter the clinical symptoms of the patient.
Serum cortisol (FC) | Week 0, Week 8
  Serum cortisol (FC) will be measured to assist in reflecting changes in participants' Yang deficiency constitution.
Serum corticosterone (CORT) | Week 0, Week 8
  Serum corticosterone (CORT) will be measured to assist in reflecting changes in participants' Yang deficiency constitution.
Serum adrenocorticotropic hormone (ACTH) | Week 0, Week 8
  Serum adrenocorticotropic hormone (ACTH) will be measured to assist in reflecting changes in participants' Yang deficiency constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Zhou, MD, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine

REFERENCES:
- [Background] Park BY, Lee MJ, Kim M, Kim SH, Park H. Structural and Functional Brain Connectivity Changes Between People With Abdominal and Non-abdominal Obesity and Their Association With Behaviors of Eating Disorders. Front Neurosci. 2018 Oct 11;12:741. doi: 10.3389/fnins.2018.00741. eCollection 2018. PMID 30364290
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Freisling H, Arnold M, Soerjomataram I, O'Doherty MG, Ordonez-Mena JM, Bamia C, Kampman E, Leitzmann M, Romieu I, Kee F, Tsilidis K, Tjonneland A, Trichopoulou A, Boffetta P, Benetou V, Bueno-de-Mesquita HBA, Huerta JM, Brenner H, Wilsgaard T, Jenab M. Comparison of general obesity and measures of body fat distribution in older adults in relation to cancer risk: meta-analysis of individual participant data of seven prospective cohorts in Europe. Br J Cancer. 2017 May 23;116(11):1486-1497. doi: 10.1038/bjc.2017.106. Epub 2017 Apr 25. PMID 28441380
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Dalle Grave R, Calugi S, El Ghoch M. Lifestyle modification in the management of obesity: achievements and challenges. Eat Weight Disord. 2013 Dec;18(4):339-49. doi: 10.1007/s40519-013-0049-4. Epub 2013 Jul 27. PMID 23893662
- [Background] Khera R, Murad MH, Chandar AK, Dulai PS, Wang Z, Prokop LJ, Loomba R, Camilleri M, Singh S. Association of Pharmacological Treatments for Obesity With Weight Loss and Adverse Events: A Systematic Review and Meta-analysis. JAMA. 2016 Jun 14;315(22):2424-34. doi: 10.1001/jama.2016.7602. PMID 27299618
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] Andersen CJ, Murphy KE, Fernandez ML. Impact of Obesity and Metabolic Syndrome on Immunity. Adv Nutr. 2016 Jan 15;7(1):66-75. doi: 10.3945/an.115.010207. Print 2016 Jan. PMID 26773015
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Sheng J, Jin X, Zhu J, Chen Y, Liu X. The Effectiveness of Acupoint Catgut Embedding Therapy for Abdominal Obesity: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Jun 23;2019:9714313. doi: 10.1155/2019/9714313. eCollection 2019. PMID 31341504